CLINICAL TRIAL: NCT05510128
Title: Evaluation of the Effectiveness of the Application of a Protocol for the Management of Female Functional Urinary Signs in French Community Pharmacies
Brief Title: Evaluation of the Effectiveness of a Protocol for the Management of Female Functional Urinary Signs
Acronym: PharmaCyst'
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A premature termination was decided following the publication of the order authorizing the pharmacist to dispense antibiotics for simple cystitis in women. Thus the experimental practice of the study joins very strongly with the new practice.
Sponsor: University Hospital, Angers (Other Government)
Collaborators: agence régionale de santé Pays de la Loire (Unknown); union régionale des professionnels de santé pharmaciens libéraux Pays de la Loire (Unknown); Direction Générale de l'offre de Soins (DGOS) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 49RC22_0240
Record Dates: First submitted 2022-07-20; First posted 2022-08-22 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cystitis Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Management with the protocol (Experimental): Patients who participate in the study in the experimental arm benefit from an adapted management, which falls under the application of the national cooperation protocol.
  This management may lead to the dispensing of an antibiotic by the pharmacist himself.
  Interventions: Other: Pharmacist management
- Standard care (No Intervention): Patients participating in the study in the control arm will benefit from a management comparable to the current one. In addition to a reminder of the hygienic and dietary rules by the pharmacist, the patient may be offered a drug indicated for improving urinary comfort.
  The pharmacist should also remind the patient that she can consult a doctor, especially in case of non relief or aggravation of symptoms.

INTERVENTIONS:
Other: Pharmacist management — When a patient comes to the pharmacy with signs of urinary burning, the following will follow:
  * Completion of the acute cystitis symptoms score (ACSS) questionnaire.
  * Measure the temperature.
  * Perform a urine dipstick.
  If the patient's temperature is normal, the urine dipstick is positive, and the absence of pain in the lumbar fossa is verified, the pharmacist can dispense an appropriate antibiotic himself. A reminder of the hygienic-dietary rules is also issued, and a communication to the patient's general practitioner will be made.
  Arms: Management with the protocol

SUMMARY:
Every year, between 4 and 6 million French people are affected by a urinary infection; the vast majority of these are women. Although the diagnosis of an uncomplicated urinary tract infection is simple to make, it requires prompt medical management to relieve the symptoms. The lack of immediate of a physician can slow down the management of patients affected by this condition, and lead to an inappropriate referral of patients to the emergency services.

Because of their wide availability, accessibility, and geographical distribution throughout the country, pharmacists are primary health care professionals who are regularly called upon to respond to patients with this type of infection.

A national protocol exists in France, but it is very difficult to apply. The PharmaCyst' study aims to evaluate its application in community pharmacies.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥ 18 and <65 years
* Patient with less than 3 days of simple urinary tract infection symptoms:

  * Burning, pain on urination
  * Dysuria
  * Pollakiuria
  * Urinary urgency
* Patient affiliated or beneficiary of a social insurance
* Patient having signed an informed consent.

Exclusion Criteria:

* More than 3 cystitis in the last 12 months;
* Last cystitis less than 15 days old;
* Presence of fever;
* Presence of back pain;
* Presence of a functional or organic anomaly of the urinary tract (bladder residue, vesico-ureteral reflux, lithiasis, tumor);
* Pruritus or vaginal discharge;
* Vomiting, diarrhea, diffuse abdominal pain;
* Risk factors for C3G-resistant enterobacteria infection (grade B):
* Exposure to an antibiotic (amoxicillin-clavulanic acid, C2G, C3G, fluoroquinolones) within the previous 3 months;
* A nosocomial or healthcare-associated infection;
* A history of colonization or infection with C3G-resistant enterobacteria within the last 3 months;
* A trip to a foreign country within the last 3 months in known geographical areas at risk (in particular the Indian subcontinent, South-East Asia, the Middle East and North Africa, the Mediterranean basin);
* Hospitalization within 3 months;
* Hospitalization within 6 months for UTI;
* Known severe renal insufficiency (creatinine clearance < 30 mL/min);
* Severe immunosuppression or immunosuppressive treatments;
* Contraindications to drugs planned for experimental management (pivmecillinam and fosfomycin) or combination of drugs not recommended;
* Pregnant women (confirmed or suspected pregnancy), breastfeeding women or women in labour;
* Person deprived of liberty by judicial or administrative decision;
* Person under forced psychiatric care;
* Person admitted to a health or social institution for purposes other than research;
* Person subject to a legal protection measure;
* A person who is unable to give consent.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender identity
Enrollment: 145 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
The evolution of the symptoms at D3 | Enrollment, Day 3
  Difference in the score from the first part of the Acute Cystitis Symptome Score questionnaire. The minimum value is 0 and the maximun value is 18. A higher score mean worse outcome

SECONDARY OUTCOMES:
The evolution of the symptoms at D10 | Enrollment, Day 10
  Difference in the score from the first part of the Acute Cystitis Symptome Score questionnaire. The minimum value is 0 and the maximun value is 18. A higher score mean worse outcome
Use of a medical consultation or an emergency service | At 3 days
  Number of consultations provided
Use of a medical consultation or an emergency service | At 10 days
  Nature of consultations provided
Performing a urine dipstick | Enrollment, Day 3, Day 10
  Number of urine dipstick performed
Performing a urine culture | At 3 days and 10 days
  Number of urine culture performed
Taking medication to relieve the symptoms of the infection | Enrollment,
  Number of medication used
Taking medication to relieve the symptoms of the infection | Day 3,
  Nature of medication used
Taking medication to relieve the symptoms of the infection | Day 10
  Nature of medication used
Occurrence of an adverse event at D3 and D10 | At 10 days
  Number of adverse events
Occurrence of an adverse event at D3 and D10 | At 3 days
  Nature of adverse events
Recurrence of a urinary tract infection within 3 months (M3) | At 3 months
  Number of cystitis encountered

OTHER OUTCOMES:
Patients' satisfaction | At 10 days
  Satisfaction measured by a Likert scale. The minimum value is 0 and the maximun value is 27. A higher score mean good outcome
Patients' care overall satisfaction | At 10 days
  Satisfaction measured by a Likert scale. The minimum value is 0 and the maximun value is 10. A higher score mean good outcome
Pharmacists' satisfaction | through study completion, an average of 12 months
  Satisfaction measured by a Likert scale. The minimum value is 0 and the maximun value is 51. A higher score mean good outcome
Pharmacists' experience | through study completion, an average of 12 months
  We will conduct semi-structured interviews with investigator pharmacyst who want's it We will explore Pharmacists' experience on the clinical research participation, including its Strengths, Weaknesses, Opportunities, and Threats.
Overall satisfaction of patients | At 10 days
  Overall satisfaction level of patients with the care provided in pharmacies. The minimum value is 0 and the maximun value is 10. A higher score mean good outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Faure, Professor, Principal Investigator — University of Angers; Aline Ramond-Roquin, Professor, Study Director — University of Angers
Locations (14):
- France (14):
  - Pharmacie du Pays De Retz, Bourgneuf-en-Retz
  - Pharmacie de Brûlon, Brûlon
  - Pharmacie Degueille, Chemazé
  - Pharmacie Nicolleau-Dilé, Chemillé-Melay
  - Pharmacie des Halles, Craon
  - Pharmacie de la Place, La Ferté-Bernard
  - Pharmacie de la Pointe, Le Mans
  - Pharmacie du Centre, Le May-sur-Èvre
  - Pharmacie du Louet, Mûrs-Erigné
  - Pharmacie des Arcades, Nozay
  - Pharmacie Deroche, Roézé-sur-Sarthe
  - Pharmacie Llacuna, Sainte-Anne-sur-Brivet
  - Pharmacie du Chemin Vert, Saumur
  - Pharmacie de la Source, Sougé-le-Ganelon

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).